CLINICAL TRIAL: NCT07175090
Title: Evaluation of the Effectiveness of a Novel Coconut Oil Mouth Rinse on Periodontal Parameters: A Randomized Controlled Trial
Brief Title: Evaluation of Coconut Oil Mouth Rinse on Periodontal Parameters
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pristina (Other)
Responsible Party: Principal Investigator, Kastriot Meqa, University assistant, University of Pristina
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 312/3
Record Dates: First submitted 2025-09-04; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-04

CONDITIONS: Periodontitis, Adult; Mouthwash
MeSH Terms: conditions — Chronic Periodontitis | interventions — Coconut Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Placebo Comparator)
  Interventions: Other: Placebo
- Group B (Active Comparator)
  Interventions: Combination Product: Coconut oil

INTERVENTIONS:
Combination Product: Coconut oil — The rinse is used three times a day during three weeks
  Arms: Group B
Other: Placebo — Inactive ingredients with same taste and colour
  Arms: Group A

SUMMARY:
This study was based on testing a new natural mouthwash with coconut oil and xylitol as active agents to a placebo rinse on new periodontal parameters

ELIGIBILITY:
Inclusion Criteria:

* Periodontitis grade I, II, III

Exclusion Criteria:

* less than 20 teeth

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Improvement of gingival appearance | Three weeks of mouthrinse use
  The gingival index will be assessed before and after mouthrinse use

SECONDARY OUTCOMES:
Gingival bleeding | Three weeks after mouthrinse use
  The presence of gingival bleeding will be assessed before and after mouthrinse use

CONTACTS AND LOCATIONS:
Locations (1):
- University of Prishtina Dentistry School, Pristina, Kosovo